CLINICAL TRIAL: NCT04842981
Title: Interleukin-6 Inhibitors and Drug-drug Interactions in Patients With Rheumatoid Arthritis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow recruitment due to COVID19.
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); King Christian X´Hospital for Rheumatic Diseases (Other); Sygehus Lillebaelt (Other); Odense Patient Data Explorative Network (Other)
Responsible Party: Principal Investigator, Ann-Cathrine Dunvald, Principal investigator, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AKF-398
Record Dates: First submitted 2021-03-23; First posted 2021-04-13 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Arthritis, Rheumatoid; Interaction
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; sarilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interleukin 6 receptor antibody (Experimental): Tocilizumab, 162 mg subcutaneous, once every week OR Sarilumab, 200 mg subcutaneous, once every two weeks.
  Interventions: Drug: Tocilizumab; Drug: Sarilumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab and Sarilumab are considered equal. Patients are assigned the treatment based on national and local guidelines. Intervention will be administered according to the approved posology.
  Other Names: RoActemra
Drug: Sarilumab — Tocilizumab and Sarilumab are considered equal. Patients are assigned the treatment based on national and local guidelines. Intervention will be administered according to the approved posology.
  Other Names: Kevzara

SUMMARY:
With this study the investigators aim to assess if drug metabolism changes in patients with rheumatoid arthritis when an interleukin (IL)-6 inhibitor is initiated.

Patients with rheumatoid arthritis have an increased level of inflammation in the body which can lead to decreased expression and activity of drug metabolizing enzymes in the liver. This will lead to a decreased metabolism and excretion of drugs. The inflammation is driven by a number of proinflammatory cytokines e.g., IL-6. The investigators hypothesize that patients with rheumatoid arthritis initiating treatment with an IL-6-receptor inhibitor (anti-IL-6R) will obtain a normalization of the activated IL-6-pathway resulting in increased expression and activity of drug metabolizing enzymes and hence increased metabolism. Ultimately, this normalization of drug metabolism could lead to insufficient efficacy of a wide variety of drugs.

The investigators will perform a clinical pharmacokinetic trial. The study will include patients with active rheumatoid arthritis and a need to initiate treatment with an IL-6 receptor antibody. Patients will ingest a 6-drug cocktail consisting of probes for specific CYP enzymes. Plasma and urine will be drawn over 6 hours to determine concentrations of the drugs and their metabolites. Patients will then initiate IL-6 receptor antibody treatment and to assess both short- and long-term impact of altered inflammation, the same 6-drug cocktail will be ingested, and concentrations measured, after three weeks and three months. To help understand the mechanism and the putative involvement of inflammation, markers of inflammation such as cytokines, transcription factors, etc. will also be assesses.

ELIGIBILITY:
Inclusion Criteria:

* Active rheumatoid arthritis
* Age 18-75 years
* eGFR > 30 mL/min
* absolute neutrophil count (ANC) ≥ 2 x 109 /L
* Platelet count > 150 x 103 /μL (corresponding to >150 x 109 /L)
* ALAT in the normal range or within 1.5x the upper limit of normal.
* Use of effective contraception (only woman of childbearing potential)
* Negative test for hepatitis and tuberculosis

Exclusion Criteria:

* Known sensitivity to any of the medications used.
* Active severe infections
* Malignancy
* Diverticulitis
* Intake of medications which can influence the safety of the patient or the results of the study. Can include prescription medications, over-the-counter medications, herbal medicines or dietary supplements. Will be assessed by the investigators.
* Participation in other clinical intervention trials.
* Pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Short-term change in CYP3A4 activity assessed by midazolam metabolic ratio. | 3 weeks
  A change in metabolic ratio of midazolam after 3 weeks of treatment with an IL-6Ra as compared to baseline. The metabolic ratio of midazolam is used to assess the activity of CYP3A4.

SECONDARY OUTCOMES:
Long-term change in CYP3A4 activity assessed by midazolam metabolic ratio. | 12 weeks
  A change in metabolic ratio of midazolam after 12 weeks of treatment with an IL-6Ra as compared to baseline. The metabolic ratio of midazolam is used to assess the activity of CYP3A4.
Short-term change in CYP1A2 activity assessed by caffeine metabolic ratio. | 3 weeks
  A change in metabolic ratio of caffeine after 3 weeks of treatment with an IL-6Ra as compared to baseline. The metabolic ratio of caffeine is used to assess the activity of CYP1A2.
Long-term change in CYP1A2 activity assessed by caffeine metabolic ratio. | 12 weeks
  A change in metabolic ratio of caffeine after 12 weeks of treatment with an IL-6Ra as compared to baseline. The metabolic ratio of caffeine is used to assess the activity of CYP1A2.
Short-term change in CYP2B6 activity assessed by efavirenz metabolic ratio. | 3 weeks
  A change in metabolic ratio of efavirenz after 3 weeks of treatment with an IL-6Ra as compared to baseline. The metabolic ratio of efavirenz is used to assess the activity of CYP2B6.
Long-term change in CYP2B6 activity assessed by efavirenz metabolic ratio. | 12 weeks
  A change in metabolic ratio of efavirenz after 12 weeks of treatment with an IL-6Ra as compared to baseline. The metabolic ratio of efavirenz is used to assess the activity of CYP2B6.
Short-term change in CYP2C9 activity assessed by losartan metabolic ratio. | 3 weeks
  A change in metabolic ratio of losartan after 3 weeks of treatment with an IL-6Ra as compared to baseline. The metabolic ratio of losartan is used to assess the activity of CYP2C9.
Long-term change in CYP2C9 activity assessed by losartan metabolic ratio. | 12 weeks
  A change in metabolic ratio of losartan after 12 weeks of treatment with an IL-6Ra as compared to baseline. The metabolic ratio of losartan is used to assess the activity of CYP2C9.
Short-term change in CYP2C19 activity assessed by omeprazole metabolic ratio. | 3 weeks
  A change in metabolic ratio of omeprazole after 3 weeks of treatment with an IL-6Ra as compared to baseline. The metabolic ratio of omeprazole is used to assess the activity of CYP2C9.
Long-term change in CYP2C19 activity assessed by omeprazole metabolic ratio. | 12 weeks
  A change in metabolic ratio of omeprazole after 12 weeks of treatment with an IL-6Ra as compared to baseline. The metabolic ratio of omeprazole is used to assess the activity of CYP2C9.
Short-term change in CYP2D6 activity assessed by metoprolol metabolic ratio. | 3 weeks
  A change in metabolic ratio of metoprolol after 3 weeks of treatment with an IL-6Ra as compared to baseline. The metabolic ratio of metoprolol is used to assess the activity of CYP2C9.
Long-term change in CYP2D6 activity assessed by metoprolol metabolic ratio. | 12 weeks
  A change in metabolic ratio of metoprolol after 12 weeks of treatment with an IL-6Ra as compared to baseline. The metabolic ratio of metoprolol is used to assess the activity of CYP2C9.

OTHER OUTCOMES:
Change in inflammation assessed by measurement of a panel of cytokines. | 3 weeks and 12 weeks
  A change in inflammation after 3 and 12 weeks of treatment with an IL-6Ra as compared to baseline. measured by a panel of inflammatory markers.

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Cathrine Dunvald, MD, Principal Investigator — University of Southern Denmark
Locations (3):
- Denmark (3):
  - Hospital South West Jutland, Esbjerg, Region Syddanmark
  - Odense University Hospital, Odense, Region Syddanmark
  - Danish Hospital for Rheumatic Diseases, Sønderborg, Region Syddanmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dunvald AD, Soltoft K, Sheetal E, Just SA, Frederiksen IEB, Nielsen F, Olsen DA, Madsen JS, Hendricks O, Stage TB. Cytochrome P450 activity in rheumatoid arthritis patients during continuous IL-6 receptor antagonist therapy. Eur J Clin Pharmacol. 2023 Dec;79(12):1687-1698. doi: 10.1007/s00228-023-03578-1. Epub 2023 Oct 13. PMID 37831074